CLINICAL TRIAL: NCT05280041
Title: An Online Self-help Intervention for Coping With the Loss of a Partner: Randomised Controlled Trial
Brief Title: Optimising an Online Self-help Program for Coping With the Loss of a Spouse
Acronym: SOLENA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jeannette Brodbeck (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor-Investigator, Jeannette Brodbeck, Professor, University of Applied Sciences and Arts Northwestern Switzerland
Organization: University of Applied Sciences and Arts Northwestern Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-02221
Record Dates: First submitted 2022-02-02; First posted 2022-03-15 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Grief
Keywords: Grief symptoms; Depression symptoms; Loneliness; Prolonged grief; Self-help online program
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: The study is a single-centered randomized control trial with three arms: Two active arms correspond to the two intervention conditions in which the content is presented in a fixed standardised order (SOLENA-F) and a self-tailored order in which the participants select the modules and their sequence (SOLENA-ST) as well as the waiting list control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fixed standardized - SOLENA-F (Experimental): In the fixed standardized arm participants will be asked to complete the study modules of the intervention (CBT intervention itself) in a fixed standardized order from module 1 to module 10. Participants will only be able to start the following module once they complete the previous one. At the beginning and at the end of each module it is emphasized what participants will do in the following module.
  Interventions: Behavioral: SOLENA - Online self-help program for older adults who lost the partner
- Self-tailored - SOLENA-ST (Experimental): In the self-tailored arm participants will be asked to complete most of the study modules of the intervention (CBT intervention itself) in a flexible format, according to their own needs at each moment. Participants will be asked to start the intervention by completing the preparatory modules (modules 1 and 2) following a fixed order. After completion of module 2, all the remaining modules become available at the same time. At the beginning and at the end of each module, participants are invited to reflect on their own needs and to complete the modules that better meet them.
  Interventions: Behavioral: SOLENA - Online self-help program for older adults who lost the partner
- Waiting list control group (No Intervention): Participants in this group will start the intervention 10 weeks after the randomization. Participants in the waiting list control group will be randomly distributed by the fixed standardised and self-tailored arms. This arm will follow the exact same procedure of the active arms.

INTERVENTIONS:
Behavioral: SOLENA - Online self-help program for older adults who lost the partner — SOLENA follows the most relevant CBT elements of interventions for prolonged grief: 1) Exposure, e.g., telling the story of the loss; 2) cognitive reappraisal or restructuring of individual dysfunctional thoughts associated with the loss; 3) integration and restoration including self-care and social reengagement; and 4) behavioural activation. SOLENA's content is provided through a conversational virtual agent, Sol, who guides the user through the Study section the CBT intervention itself. In 10 study modules that address either the acceptance of the loss or the restoration and adaptation to a new life, SOLENA includes 1) readings, i.e., texts based about grief related topics that provide the background and rational for the module; and 2) exercises to encourage mourners to actively reflect on their grief and apply their new knowledge to their daily life and to practise the new routines regularly. SOLENA also provides users with the Notebook, Activities, and My Support sections.
  Other Names: SOLENA
  Arms: Fixed standardized - SOLENA-F; Self-tailored - SOLENA-ST

SUMMARY:
When someone has lost his or her partner, feelings of grief are normal and usually diminish over time. However, for some people, strong feelings of grief persist. For coping with grief, it is important to learn to accept the loss, experience the pain of grief, adjust to an environment without the deceased person, and withdraw emotional energy and focus it on other relationships. Loss-oriented tasks, such as grief work, and restoration-oriented tasks, such as attending to life changes, engaging in new activities and finding new roles and identities, are both essential.

The program is designed to be completed in 10 weeks and recommends that mourners complete one module or topic a week. To examine the benefits of SOLENA, this study will compare the answers of mourners that completed the intervention with the mourners of the control group, which will wait to complete the intervention. The group that completed the intervention is divided in two sub-groups. One group of mourners will complete the intervention in a fixed order, while the other will complete it in a self-tailored order according to their own needs at each moment. Specifically, the study examines how well the self-help program reduces grief, depression symptoms, and loneliness and examines whether the topics of the study modules are presented in a given order or whether participants can work on the topics according to their current needs makes a difference. Ultimately, it is expected that the self-tailored version leads to more benefits than completing SOLENA's modules in a fixed order.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE

The death of a spouse is a frequent and very stressful critical life event in later life. The loss of a partner involves the adaptation of daily routines which can be even more challenging when social, physical, and financial resources decline in later life. Grief and psychological distress after the loss of a spouse are normative reactions. For most people, grief intensity weakens to a manageable degree within several weeks or months. However, some individuals are less able to cope with bereavement and show symptoms of disturbed or prolonged grief or adaptation problems.

To support coping with the loss of a significant person, the Task model identifies four tasks of mourning, namely accepting the reality of the loss, experiencing the pain of grief, adjusting to an environment without the deceased person, and withdrawing emotional energy and reinvesting it in another relationship. Moreover, the dual-process model of coping with bereavement posits that a dynamic coping process oscillating between loss-oriented tasks such as grief work and restoration-oriented tasks such as attending to life changes is essential for adjustment.

Based in these two models, Brodbeck and colleagues developed LIVIA, a text-based self-help online program to support the loss of the spouse, which has proved its efficacy for mourning older adults from a general population. LIVIA is rooted in cognitive behavioural therapy, including the most relevant treatment elements to support the mourning process: exposure, cognitive reappraisal, integration, and restoration as well as self-care and social reengagement treatment components.

LIVIA confirmed that the intervention is also efficacious for milder grief symptoms. Compared to the control group, the intervention resulted in significant reductions in grief (d = 0.81), depression (d = 0.59), psychopathological distress (d = 0.39) (primary outcomes), embitterment (d = 0.37), loneliness (d = 0.37) and an increase in life satisfaction (d = -0.41) (secondary outcomes). These gains were maintained over three months. Improvements were similar among participants with low, medium, or high levels of grief at baseline. Therefore, LIVIA provides a promising basis for the development of a more sophisticated and attractive intervention with a more inclusive target group, e.g., mourners of all ages who lost their spouse within the previous six months, while still seeking help for coping with the loss.

Apart from extending the target population of the intervention, SOLENA also aims to examine whether the efficacy of LIVIA can be increased by providing a self-tailored version, in which the users can chose the content that is relevant for them and that best fits their current needs.

MAIN HYPOTHESES

Primary outcome: Grief

1. Efficacy of SOLENA: It is hypothesized that SOLENA will decrease grief significantly compared to the waiting list control group.
2. Stability of the effects: It is hypothesized that SOLENA leads to stable effects on grief across 10 weeks.
3. Comparison of the two active arms: When assessing the presentation format of SOLENA, it is hypothesized that self-tailored arm will lead to higher decrease of grief than the standardised arm.

   Secondary outcomes: Depression symptoms and perceived loneliness
4. Efficacy of SOLENA: It is hypothesized that SOLENA will decrease depression symptoms and perceived loneliness significantly compared to the waiting list control or treatment as usual group.
5. Stability of the effects: It is hypothesized that SOLENA leads to stable effects on depression symptoms and loneliness across 10 weeks.
6. Comparison of the two active arms: When assessing the presentation format of SOLENA, it is hypothesized that self-tailored arm will lead to higher depression symptoms and loneliness than the standardised arm (superiority hypothesis).

RECRUITMENT AND PROCEDURE

Recruitment of participants will be conducted via newspaper articles, social media, internet forums, and personal contacts to healthcare workers and churches. Potential participants will find a description of the study and the intervention on the project website, from where they can register at the study. All potential participants can contact the study management to ask questions or clear eventual doubts about the study. This presentation is compiled in accordance with the general guidelines for clinical trials published by the Swiss Ethics Committees on research involving humans for the creation of an informed consent form (ICF) for information transfer.

After receiving adequate and sufficient information about the study, the participants will declare consent by signing the ICF. All participants must confirm to have read this information before being allowed to participate in the study.

After sending back the signed informed consent, participants will be invited to fill out the baseline measures on REDCap and take part in a short telephone call for screening the inclusion and exclusion criteria.

Participants will be randomised to one of the three study arms (fixed-standardized, self-tailored or waiting list control group) and will receive the participant code to connect their data with study condition, ensuring confidentiality and privacy.

For 10 weeks, starting at t0, participants will be asked to use the text-based program, SOLENA, to support their grief process and to complete the working alliance (goal & task), change mechanisms measures, and the self-check mood monitoring.

At week 10 (t1, post-intervention), participants of the active arms will be asked to complete the primary and secondary measures. At this moment, the waiting-list control group starts using SOLENA and complete baseline measures.

At week 20 (t2, follow-up), participants of the active arms will be asked to complete primary and secondary outcome measures to assess stability of program's effects. Also at this time, participants in the waiting list control group will complete post-intervention measures.

At week 30 (t3), participants in the waiting list control group will complete follow-up measures.

STATISTICAL ANALYSES PLAN

Statistical analyses

Analyses will be conducted according to the intention-to-treat paradigm. Linear mixed-models, which will be used in this study, allow a different number of measurement points per participants and are thus less sensitive to missing data. Time will be included (pre vs post intervention measures and post intervention vs follow-up measures), group (self-tailored and standardised vs. waiting list control condition) and interaction terms as predictors of the outcome variables. Cohens d will be calculated as effect size for all observed outcome variables. To analyse the longitudinal interplay of predictor and mediator variables, path analyses will be conducted. Analyses will be conducted in SPSS, R and Mplus. Any deviation from the original statistical plan will be described and justified in the final trial report. There are no statistical stopping rules in this trial.

SAMPLE SIZE CALCULATIONS

The study is mainly powered for the efficacy and stability hypotheses, i.e., the main and interaction effects of the active conditions compared to the waiting list control on the reduction of grief, depression symptoms, and loneliness. The sample size needed was obtained conducting a power analysis with a probability level of .05 and a power of 0.80 with G*Power based on the results of the evaluation of LIVIA, i.e., large to moderate effects.

For the comparison of SOLENA and a waiting list condition, it is expected a large effect size of d > .80 or f > .4. For the comparison of the standardised and the self-tailored arms, it is expected a small to moderate effect between f = .25 and .15 in favour of the self-tailored arm. Figure 4 presents the power analyses for a repeated measures ANOVA with a within-between interaction for three groups.

A minimum of 85 participants will be included, with an allocation ratio of 35:35:15 for the two active conditions and the waiting list control group. There is no statistical criterion for terminating the trial as more than 85 participants allow more sophisticated moderator analyses for example regarding the time since the loss.

Data collection and analysis

Data are assessed using online questionnaires programmed in REDCap. Data integrity is enforced through a variety of mechanisms, i.e., referential data rules, valid values, range checks, and consistency checks. The option to choose a value from a list of valid codes and a description of what each code means is available where applicable. Checks are applied at the time of data entry into a specific field. In addition, data on the use of the self-help sessions are collected within the platform. All data will be saved in an anonymous way only identified by a code which is not related to the participant's identity. Servers are protected by high-end firewall systems. Only the researchers directly involved in the study have access to the data.

Handling of missing data and drop-outs

Dropout are defined as participants who withdraw actively from the intervention after randomisation or who do not fill out the post-intervention in spite of two reminders. As for missing data, by withdrawing actively from the intervention, an e-mail will be sent with a REDCap link to the respective participants asking them to complete the post and follow-up questionnaires, nonetheless, thereby enabling us to conduct intention-to-treat analyses. In any case, all drop-outs are a part of the intent-to-treat sample as they have been randomised and are included in the analyses. Analyses of the extent of missing data will be conducted to explore the missing data patterns and determine the type of missing data (Missing Completely at Random, Missing at Random, Not Missing at Random). Missing values will be substituted using multiple imputations. Sensitivity analyses will explore the impact of the imputation of missing values.

ELIGIBILITY:
Inclusion Criteria:

* Experience of spousal bereavement
* Seeking help for coping with grief or the psychosocial adaptation to a life without the partner
* Having access to an internet connection and adequate equipment
* Mastery of the German language
* An informed consent by the participant.

Exclusion Criteria:

* Loss less than one month ago
* Acute suicidality
* Inability to follow the procedures of the study, e.g., due to comprehension problems, visual impairment, lack of sufficient motor skills or severe psychological or somatic disorders which require immediate treatment which impedes the continuous work on the self-help programme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2025-12-17 (Actual); Study Completion 2025-12-18 (Actual)

PRIMARY OUTCOMES:
Grief: Texas Revised Inventory of Grief - German Version | At week 10 (post-intervention)
  Grief is assessed with the Texas Revised Inventory of Grief - German Version. The TRIG is a widely used measure to assess the severity of grief. The TRIG German version is a 16-item measure to assess the severity of grief from 1 = completely true to 5 = completely false. The scale ranges from 1 to 80, higher values indicate higher levels of grief.

SECONDARY OUTCOMES:
Depression symptoms measured by The Patient Health Questionnaire (PHQ-9) German version. | At week 10 (post-intervention)
  Depression symptoms will be measured by the Patient Health Questionnaire (PHQ-9). The PHQ-9 corresponds to the depression assessment module, which scores each of the nine diagnostic criteria for major depression in Diagnostic and Statistical Manual Fourth Edition. For each item, answer format is a scale from '0' (not at all) to '3' (nearly every day). The scale ranges from 0 to 27, higher values indicate higher levels of depression.
Perceived loneliness measured by the Jong Gierveld Loneliness Scale | At week 10 (post-intervention)
  Perceived loneliness will be measured with the de Jong Gierveld Loneliness Scale. This will use the revised and shortened version of the scale that 6 items that resolve into social and emotional subscales. The items can be answered on a 5-point scale from '1' (yes) to '5' (no). The scale ranges from 1 to 30, higher values indicate lower levels of loneliness.

OTHER OUTCOMES:
User satisfaction with the program, measured by Patient Satisfaction Questionnaire (ZUF-8) | At week 10 (post-intervention)
  The ZUF-8 is a self-report measure that explores patients' overall satisfaction with the treatment. It contains eight items that are rated on a 4-point scale from 1 - low satisfaction to 4 - high satisfaction. The scale ranges from 1 to 32, higher values indicate higher satisfaction. The instrument was adapted to explore patients' satisfaction with the particular Internet intervention studied in this trial.
Stability of improvement in grief: Texas Revised Inventory of Grief - German Version | At week 20 (follow-up of the intervention)
  Grief is assessed with the Texas Revised Inventory of Grief - German Version . The TRIG is a widely used measure to assess the severity of grief. The TRIG German version is a 16-item measure to assess the severity of grief from 1 = completely true to 5 = completely false. The scale ranges from 1 to 80, higher values indicate higher levels of grief.
Stability of improvement in depression symptoms measured by The Patient Health Questionnaire (PHQ-9) German version. | At week 20 (follow-up of the intervention)
  Depression symptoms will be measured by the Patient Health Questionnaire (PHQ-9). The PHQ-9 corresponds to the depression assessment module, which scores each of the nine diagnostic criteria for major depression in Diagnostic and Statistical Manual Fourth Edition. For each item, answer format is a scale from '0' (not at all) to '3' (nearly every day). The scale ranges from 0 to 27, higher values indicate higher levels of depression.
Stability of improvement in perceived loneliness measured by the Jong Gierveld Loneliness Scale | At week 20 (follow-up of the intervention)
  Perceived loneliness will be measured with the de Jong Gierveld Loneliness Scale. This will use the revised and shortened version of the scale that 6 items that resolve into social and emotional subscales. The items can be answered on a 5-point scale from '1' (yes) to '5' (no). The scale ranges from 1 to 30, higher values indicate lower levels of loneliness.
Possible change mechanisms assessed with a 5-item short version based on the Bern patient questionnaire | Through intervention completion, from week 1 to week 10.
  Session outcomes as possible change mechanisms are assessed with a 5-item short version based on the Bern patient questionnaire, including the rating of the overall helpfulness of the module and the matching of participant's needs and presented content, as well as gains in self-esteem, mastery experiences, and insight. Participants will be asked to complete the session outcomes items (Self-reflection survey) after the completion of each submodule and module. The items are rated on a scale ranging from -3 to 3 (not at all; no; rather not; neither; rather yes; yes; yes, exactly). The items can be answered on a 5-point scale from '1' (yes) to '5' (no). The scale ranges from -15 to 15, higher values indicate more improvement.
Working alliance during the intervention, Goals and Task scale | Week 3, week 6 and week 9 of the intervention
  The working alliance inventory (WAI), is a measure of the therapeutic alliance, a key variable that accounts for treatment outcomes and clients' satisfaction across interventions. The items of the WAI-I were derived from the WAI-SR. We will use the subscale, Task & Goals (T&G) that measures user's agreement with tasks and goals of program. Items are rated on a 5-point Likert scale ranging from 1 = 'never' to 5 = 'always'. The items can be answered on a 5-point scale from '1' (yes) to '5' (no). The scale ranges from 1 to 40, higher values indicate a better working alliance.

CONTACTS AND LOCATIONS:
Overall Officials: Jeannette Brodbeck, PhD, Principal Investigator — University of Applied Sciences and Arts Northwestern Switzerland
Locations (1):
- University of Applied Science Northwestern Switzerland, Olten, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brodbeck J, Berger T, Znoj HJ. An internet-based self-help intervention for older adults after marital bereavement, separation or divorce: study protocol for a randomized controlled trial. Trials. 2017 Jan 13;18(1):21. doi: 10.1186/s13063-016-1759-5. PMID 28086836
- [Background] Brodbeck J, Berger T, Biesold N, Rockstroh F, Znoj HJ. Evaluation of a guided internet-based self-help intervention for older adults after spousal bereavement or separation/divorce: A randomised controlled trial. J Affect Disord. 2019 Jun 1;252:440-449. doi: 10.1016/j.jad.2019.04.008. Epub 2019 Apr 8. PMID 31003114
- [Background] Aoun SM, Breen LJ, Howting DA, Rumbold B, McNamara B, Hegney D. Who needs bereavement support? A population based survey of bereavement risk and support need. PLoS One. 2015 Mar 26;10(3):e0121101. doi: 10.1371/journal.pone.0121101. eCollection 2015. PMID 25811912
- [Background] Boelen PA, de Keijser J, van den Hout MA, van den Bout J. Treatment of complicated grief: a comparison between cognitive-behavioral therapy and supportive counseling. J Consult Clin Psychol. 2007 Apr;75(2):277-84. doi: 10.1037/0022-006X.75.2.277. PMID 17469885
- [Background] Eisma MC, Boelen PA, van den Bout J, Stroebe W, Schut HA, Lancee J, Stroebe MS. Internet-Based Exposure and Behavioral Activation for Complicated Grief and Rumination: A Randomized Controlled Trial. Behav Ther. 2015 Nov;46(6):729-48. doi: 10.1016/j.beth.2015.05.007. Epub 2015 May 28. PMID 26520217
- [Background] Futterman A, Holland JM, Brown PJ, Thompson LW, Gallagher-Thompson D. Factorial validity of the Texas Revised Inventory of Grief-Present scale among bereaved older adults. Psychol Assess. 2010 Sep;22(3):675-87. doi: 10.1037/a0019914. PMID 20822280
- [Background] Gomez Penedo JM, Berger T, Grosse Holtforth M, Krieger T, Schroder J, Hohagen F, Meyer B, Moritz S, Klein JP. The Working Alliance Inventory for guided Internet interventions (WAI-I). J Clin Psychol. 2020 Jun;76(6):973-986. doi: 10.1002/jclp.22823. Epub 2019 Jun 25. PMID 31240727
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Martin A, Rief W, Klaiberg A, Braehler E. Validity of the Brief Patient Health Questionnaire Mood Scale (PHQ-9) in the general population. Gen Hosp Psychiatry. 2006 Jan-Feb;28(1):71-7. doi: 10.1016/j.genhosppsych.2005.07.003. PMID 16377369
- [Background] Shear K, Frank E, Houck PR, Reynolds CF 3rd. Treatment of complicated grief: a randomized controlled trial. JAMA. 2005 Jun 1;293(21):2601-8. doi: 10.1001/jama.293.21.2601. PMID 15928281
- [Background] Stroebe M, Schut H. The dual process model of coping with bereavement: rationale and description. Death Stud. 1999 Apr-May;23(3):197-224. doi: 10.1080/074811899201046. PMID 10848151
- [Derived] Brodbeck J, Jacinto S, Gouveia A, Mendonca N, Madorin S, Brandl L, Schokking L, Rodrigues AM, Goncalves J, Mooser B, Marques MM, Isaac J, Nogueira V, Matos Pires A, van Velsen L. A Web-Based Self-help Intervention for Coping With the Loss of a Partner: Protocol for Randomized Controlled Trials in 3 Countries. JMIR Res Protoc. 2022 Nov 30;11(11):e37827. doi: 10.2196/37827. PMID 36449341